CLINICAL TRIAL: NCT06842784
Title: Impact of Extreme Heat on Myocardial Blood Flow and Flow Reserve in Young and Older Adults
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The American Society of Echocardiography (Unknown)
Responsible Party: Principal Investigator, James MacNamara, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU_2019_1759_MCE; 1R01AG069005 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Aging; Heat Stress; Hyperthermia; Heat Strain
MeSH Terms: conditions — Heat Stress Disorders; Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young participants: Individuals aged 18-39 years
  Interventions: Other: Ambient heat stress
- Older participants: Individuals aged 65 years or older
  Interventions: Other: Ambient heat stress

INTERVENTIONS:
Other: Ambient heat stress — 3-hour ambient heating in 44°C and 20% relative humidity

SUMMARY:
Extreme heat causes a disproportionate number of hospitalizations and deaths in older adults relative to any other age group. Importantly, many hospitalizations and deaths are primarily due to cardiovascular events such as myocardial infarction. Previous data indicate that older adults have attenuated skin blood flow and sweating responses when exposed to heat, resulting greater increase in core body temperature. Despite these observations, relatively little is known about the risk for myocardial ischemia potentially contributing to the aforementioned higher morbidity and mortality in older adults during heat waves. The broad objective of this work is to determine the impact of ambient heat exposure on myocardial blood flow and flow reserve in young and older adults. Aim 1 will test the hypothesis that older adults exhibit attenuated myocardial flow reserve compared to young adults during heat stress. Aim 2 will determine if the percent of maximal myocardial flow reserve (assess via vasodilator stress) during heat exposure is higher in older adults compared to young adults. The expected outcome from this body of work will improve our understanding of the consequences of aging on cardiovascular responses to ambient heat stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female individuals
* 18-35 years or 65+ years of age
* Free of any underlying moderate to serious medical conditions

Exclusion Criteria:

* Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, uncontrolled hypertension, and uncontrolled hypercholesterolemia.
* Taking of any medications (such as beta blockers and non-dihydropyridine calcium channel blockers) that have known influences on either cardiac function or sweating responses.
* Abnormalities detected on routine screening.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2
* Pregnant individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be healthy younger and older individuals identified from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial flow reserve | The difference in the change from baseline to a vasodilator stress test and the change from baseline to after 3-hours of heat stress.
  Measured via myocardial contrast echocardiography.
Myocardial blood flow | The change from baseline to after 3 hours of heat stress.
  Measured via myocardial contrast echocardiography.

SECONDARY OUTCOMES:
Core temperature | The change from baseline to after 3 hours of heat stress..
  Measured via ingestible telemetric pill.
Indices of left and right ventricular function | At baseline and after 3 hours of heat stress.
  Measured via echocardiography.
Heart rate | At baseline, during exercise- after 20 minutes and 2 hours in the heat, and at rest after 3 hours of heat stress.
  Measured via electrocardiogram.
Blood pressure | At baseline, during exercise- after 20 minutes and 2 hours in the heat, and at rest after 3 hours of heat stress.
  Measured via automated auscultation of the brachial artery.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No